CLINICAL TRIAL: NCT04286828
Title: An Investigation of Knee Position Sense, Balance, and Dual Task Performance in Different Phases of Menstrual Cycle in Females With Multiple Sclerosis
Brief Title: Position Sense, Balance, and Dual Task Performance at the Menstrual Cycle in Females With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-17
Record Dates: First submitted 2020-02-23; First posted 2020-02-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis; Neurologic Symptoms; Menstrual Cycle
Keywords: Multiple Sclerosis; Proprioception; Postural balance; Task performance and analysis
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations | interventions — Proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females with Multiple Sclerosis: Patients with confirmed diagnosis of clinically definite MS and physician-administered EDSS range of 1-3.5.
  Interventions: Other: Position Sense; Other: Balance; Other: Dual Task Performance
- Healthy Females: 20 healthy volunteers with matching ages and genders.
  Interventions: Other: Position Sense; Other: Balance; Other: Dual Task Performance

INTERVENTIONS:
Other: Position Sense — Knee position sense was evaluated with a Acumar dual digital inclinometer. Each participant was asked to wear shorts and to lie down in supine position treatment table. The lower extremity of the participant was positioned in neutral for the knee flexion movement. The placement of the digital inclinometer's attachment was the lateral ridge of the femur and tibia. We actively assisted the participant's knee to the target angle and asked the participant to hold it there for 5 seconds before returning the knee to the starting position. After returning to the starting position, participants attempted to repeat the previously attained angle. Participants indicated verbally when they felt they had reached the angle and held their position. This procedure was repeated 3 times for each limb (non-dominant and dominant). We measured the absolute difference between the target angle and the observed angle and calculated the absolute error score by averaging the 3 trials.
Other: Balance — To measure postural stability and Limits of Stability this study used a balance device, the Biodex Balance System.
  Postural Stability: The participants were focused on a characteristic dot (COP, centre of pressure) on the monitor screen. The participant's task was to balance the body in such a way that the dot was in the centre of a circle displayed on the monitor at the point of intersection of the coordinate axes. Test consisted of three 20-second trials, each separated by 10-second breaks. Measurements were repeated three times while their eyes were open/close and analyzed by calculating the average value of measurements.
  Limits of Stability: The participants are asked to complete the directional tasks displayed on a screen as quickly as possible, with the directions displayed at random. A total of 3 tests were performed, at intervals of 10 s.
Other: Dual Task Performance — The timed up and go test (TUG) was used in the evaluation of dual task performance. For this test, participants were seated on a standard armless chair and a cone was placed 3 meters away from the chair. Participants were instructed to stand up and (1) walk towards the cone, (2) turn around the cone, (3) walk back to the chair, and (4) sit back on the chair. It was stated that patients should walk without running but as fast as possible. TUG test was performed initially without task, and then with cognitive and motor tasks, respectively. Cognitive task given during the test is counting three backwards from 100 or counting the names starting with the letter "A", and motor task given is to carry three glasses of water on a tray. The time elapses between standing up from the chair and sitting back to chair was recorded as the test result. As time increases, dual task performance decreases.

SUMMARY:
The aim of this study was to investigation of knee position sense, balance, and dual task performance in different phases of menstrual cycle in females with multiple sclerosis.

Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) affecting young people and leading to demyelination and neurodegeneration. MS affects females more than males with a ratio approximately of 3:1. Important gender differences in progression and inflammatory activity of disease have been observed. Sex hormones have been thought to play an important role in this condition. It is worth noting however that sex hormones not only affect reproduction (menses/pregnancy), they also have direct effects on the nervous and immune system. In the neurologic group, especially in MS patients, it is well known that disease activity, course, and symptoms can be influenced by hormonal fluctuations in different phases of the menstrual cycle. Previous studies have reported that the variation of estrogen and progesterone during the menstrual cycle may have an effect on several neurological functions. However, these studies are mostly subjective, in the form of patient reports and in limited numbers. Smith and Studd reported that there was a premenstrual increase in disease severity as changes in the Th-1 / Th-2 balance occurred in association with decreased circulating estrogen. Withdrawal of hormones from damaged tissues that affect axonal conduction can explain the change in disease activity, course symptoms during the menstrual cycle in female with MS.

For all these reasons,investigators think that different phases of menstrual cycle change position sense, balance, and dual task performance in females with MS. Considering hormonal fluctuations occurring in the menstrual cycle, is an important criterion for organizing the rehabilitation program and evaluation in terms of physiotherapy.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effect of hormonal changes on knee position sense, balance and dual task performance throughout the menstrual cycle in females with MS.

14 females with MS and 13 healthy females with matching ages and genders were included the study. A neurologic examination was performed using the EDSS by a neurologist.

Position sense was measured with Acumar dual digital inclinometer (Acu360, Acumar, Lafayette, USA). Balance was measured with Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA). Dual task performance was evaluated with Time Up and Go test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of the MS group were as follows: patients with a confirmed diagnosis of clinically definite MS, physician-administered Expanded Disability Status Scale (EDSS) range of 1-3.5, and having regular menstrual cycle (between 21-35 days).
* Inclusion criteria of the control group were having regular menstrual cycle, and not having neurological problem, any lower extremity orthopedic problems and no use of any contraceptive agents

Exclusion Criteria:

* The exclusion criteria were: patients with acute attacks (three months prior to the study), a Mini-Mental State Examination (MMSE) score of less than 25 points, take oral contraceptive agents, and a history of orthopedic lower extremity problems or other neurological disorders.

Ages: 26 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: having regular menstrual cycle females with MS and healthy females
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Knee position sense | through study completion, an average of 1 year
  Knee position sense was evaluated with a Acumar dual digital inclinometer.The absolute error scores (in degrees) for knee flexion at 60° was calculated. As absolute error score increases, position sense decreases.
Balance | through study completion, an average of 1 year
  To measure postural stability and Limits of Stability this study used a balance device, the Biodex Balance System.
  Postural Stability: Test consisted of three 20-second trials, each separated by 10-second breaks. Measurements were repeated three times while their eyes were open/close and analyzed by calculating the average value of measurements [30]. As a result, overall stability indexes were taken into account for measurement purposes. For these indexes, a low value indicated high postural stability.
  Limits of Stability: The participants are asked to complete the directional tasks displayed on a screen as quickly as possible, with the directions displayed at random. A total of 3 tests were performed, at intervals of 10 second. The test results were used to determine a total score. The higher the total score, the better the ability of the subjects to transfer the centre of gravity.
Dual Task Performance | through study completion, an average of 1 year
  The timed up and go test was used in the evaluation of dual task performance. Timed up and go test was performed initially without task, and then with cognitive and motor tasks, respectively. Cognitive task given during the test is counting three backwards from 100 or counting the names starting with the letter "A", and motor task given is to carry three glasses of water on a tray. The time elapses between standing up from the chair and sitting back to chair was recorded as the test result. As time increases, dual task performance decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)